CLINICAL TRIAL: NCT02650141
Title: Efficacy of Experienced Chinese Herbal Formulas for the Treatment of Different Types of Precocious Puberty: A Single-blinded Randomized Controlled Trial
Brief Title: Clinical Trial of Experienced Chinese Herbal Formulas on Different Types of Precocious Puberty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jian Yu, Professor, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO.12401905505
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ziyinxiehuo Granules (Experimental): Children of ziyinxiehuo granules group will be treated with chinese herbal granules,3 times a day, for 6 months.
  Interventions: Drug: ziyinxiehuo Granules
- zishenqinggan Granules (Active Comparator): Children of zishenqinggan granules group will be treated with chinese herbal granules, 3 times a day, for 6 months.
  Interventions: Drug: zishenqinggan Granules

INTERVENTIONS:
Drug: ziyinxiehuo Granules — Ziyinxiehuo granules Herbs (1 bag ): shengdi 5g, xuanshen 3g, zexie 3g, zhimu3g, huangpai 3g, zhiguiban 2g, maiya 6g,tiandong 3g, zhigancao 2g Therapeutic Principle: Nourishing "Yin", removing "Fire" Usage: administered after dissolved, 3 times per day after breakfast and supper
  Other Names: nourishing"Yin"-removing"Fire" Granules
  Arms: ziyinxiehuo Granules
Drug: zishenqinggan Granules — Zishenqinggan granules Herbs (1 bag ): Shengdi 5g, baishao 3g, huangqin 3g, fuling 4g, danpi 3g, maiya 6g, shanzha 3g, zhebei 3g, zhigancao 2g Therapeutic Principle: replenishing "Kidney", Clearing "Liver" Usage: administered after dissolved, 3 times per day after breakfast and supper
  Other Names: replenishing "Kidney"-Clearing "Liver" Granules
  Arms: zishenqinggan Granules

SUMMARY:
Due to various complex factors, the incidence of precocious puberty is increasing rapidly. It severely threatens physical and mental health of children. It's urgent to explore effective ways to control the disease.

DETAILED DESCRIPTION:
In the research, 138 precocious puberty children are randomly divided into the Ziyinxiehuo granules group (69 cases) and Zishenqinggan granules group(69 cases). Patients in Ziyinxiehuo granules group are treated with a series of experienced chinese herbal formulas, whereas the Zishenqinggan granules group received with different series of experienced chinese herbal formulas.

ELIGIBILITY:
1. In the partial precocious puberty children：

   Inclusion Criteria:
   * Girls are diagnosed as simple early breast development, and their age of onset is less than 8 years
   * Tanner stages of breast in female patients are Tanner II and Tanner III, Diameter of mammary nucleus is less than 3cm；
   * B-type ultrasonography: the size and volume of uterus and follicle is in the normal range at the same age；
   * bone age: the bone age in the patients are the same with their actual age.

   Exclusion Criteria:
   * the bone age is advanced by more than 1 standard deviations for chronological age
   * pseudo sexual precocity, including gonadal tumor,adrenal disease,exogenous intake induced with hormone drugs or food and multiple bone fiber structure dysplasia of precocious puberty (McCune Albright syndrome)
   * heterosexual precocious puberty
2. In the mild true precocious puberty children：

Inclusion Criteria:

* Girls are diagnosed as Idiopathic central precocious puberty，and their age of onset ≤8 years
* Tanner stages of brest in female patients ≤ Tanner III stage，diameter of mammillary nucleus < 3cm
* B-type ultrasonography: the volume of uterus≥1~3ml，the diameter of follicle≥4mm;or the length of uterus ≥3.4-4cm
* bone age: compared the actual age ,the bone age is no more than 1 year and the bone age <10 years old;
* in master single test: LH >3 IU/L
* GnRH stimulation test: LH/FSH>0.6, the Peak LH 3.5~5.0 IU/L, the Peak LH 3.5~5.0 IU/L.

Exclusion Criteria:

* The central nervous system organic diseases caused sexual precocity
* congenital thyroid function reduce disease with precocious puberty, congenital adrenal hyperplasia, adrenal tumor
* ovarian or testicular neoplasms,
* McCune Albright syndrome (precocious puberty with polyostotic fibrous dysplasia and skin pigment abnormalities, pigmentation)
* there is a family history of diseases such as tumor, leukemia, diabetes, systemic lupus erythematosus, etc
* precocious puberty and partial precocious puberty

Max Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in some index of B type ultrasonography ( uterus,ovary,follicle ) | 3 months, 6months
  The investigators will measure the change of some index of B type ultrasonography ( the volume of uterus and ovary, the biggest follicle diameter )

SECONDARY OUTCOMES:
change in the mammary nucleus index | 3 months, 6 months
  The investigators will measure the change of the mammary nucleus index by the mammary diameter
change in the cumulative score of traditional Chinese medicine syndromes | 3 months, 6 months
  The investigators will measure the change in scores of chinese medicine symptoms according to the Traditional Chinese Medicine Guideline Scale: 0 - 3. 0 = None. 1 = Mild. 2 = Moderate. 3= Severe

CONTACTS AND LOCATIONS:
Overall Officials: Jian Y Jian, professor, Study Chair — Children Hospital of Fudan University
Locations (1):
- Department of Chinses Traditional Medcine； Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data will be used by the research group only.

REFERENCES:
- [Result] Sun W, Han X, Wang Y, Yu J, Yan W, Zhao J, Chen W, Xue Z. Effectiveness of ZiYin Xiehuo granules and Zishen Qinggan granules on partial precocious puberty in girls: a multicenter, randomized, single-blind, controlled trial. J Tradit Chin Med. 2018 Oct;38(5):740-745. PMID 32185991